CLINICAL TRIAL: NCT01658540
Title: Safety and Efficacy of the Drug Eluting Balloon (DEB) for the Treatment of the Superficial Femoral Artery (SFA) Ischemic Vascular Disease in Symptomatic Patients Presenting With Long Lesions: a Pilot Study
Brief Title: Drug Eluting Balloon (DEB) and Long Lesions of Superficial Femoral Artery (SFA) Ischemic Vascular Disease
Acronym: DEB-SFA-LONG
Status: Completed | Type: Observational
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO09
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Peripheral Artery Disease
Keywords: Drug Eluting Balloon (DEB) technology; long SFA lesions disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to assess safety and efficacy of the Drug Eluting Balloon (DEB) technology for the treatment of the Superficial Femoral Artery (SFA) ischemic obstructive vascular disease in patients presenting with long lesions. As secondary aim this study is going to explore treatment effect on a number of procedural and clinical endpoints in order to collect information to design a future comparative effectiveness study.

DETAILED DESCRIPTION:
The study is aimed at collecting preliminary safety and efficacy data related to the use of Drug Eluting Balloon (DEB) technology for the treatment of symptomatic Superficial Femoral Artery (SFA) ischemic vascular disease in patients presenting with long lesions.

The present clinical evaluation is intended as a prospective observational data collection of patient treatment in full accordance with institution standard practice and utilizing an approved (CE marked) DEB currently available on the market.

ELIGIBILITY:
Inclusion Criteria:

* Documented ischemic, symptomatic arterial disease in the femoral-popliteal arteries according to Rutherford Category 2, 3 or 4;
* Target lesion consists of a single solitary or multiple adjacent de novo or restenotic lesions (non-in-stent) with diameter stenosis ≥ 70% by visual estimate and cumulative lesion length ≥ 15 cm;
* Target vessel is the superficial femoral artery and/or proximal popliteal artery (above the knee);
* Life expectancy >1 year in the Investigator's opinion;
* Written informed consent.

Exclusion criteria:

Given the observational nature of the study, no study-specific but only clinical exclusion criteria will apply:

* Patient unwilling or unlikely to comply with FU schedule;
* Administration of local or systemic thrombolytic therapy within 48 hours prior to the index procedure;
* Known allergies or sensitivities to heparin, aspirin, other anticoagulant/antiplatelet therapies, and/or paclitaxel;
* Additional planned cardiac or peripheral percutaneous or surgical intervention including CABG within 30 days following the study procedure;

  * 15 cm long inflow lesion (≥50% DS) or occlusion (any length) in the ipsilateral Iliac artery;
* Failure to successfully treat < 15 cm long inflow lesion in the ipsilateral Iliac artery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by lower extremities artery disease (LEAD) and referred to the participating centres for the endovascular treatment of de novo or restenotic lesions (no in stent restenosis) in the superficial femoral and proximal popliteal arteries will be considered for the study
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
rate of primary patency | within the first 12 months after percutaneous treatment
  Primary patency is defined as freedom from the combined endpoints of clinically-driven target lesion revascularization (TLR) and >50% restenosis in the treated lesion. Clinically driven TLR is defined as any re-intervention within the target lesion due to symptoms or drop of ABI of ≥20% or >0.15 when compared to post-procedure. Restenosis > 50% is defined by a peak systolic velocity ratio (PSVR) > 2.4.

SECONDARY OUTCOMES:
composite of all Major Adverse Events (MAE) | within the first 24 months after percutaneous treatment
  evaluate the incidence of the composite of all Major Adverse Events (MAE) through 24 months i.e. the first occurrence of any of the following: death from any cause, major target limb amputation, thrombosis at the target lesion site
incidence of Major Adverse Cardiac and Cerebrovascular event (MACCE) | within the first 24 months after percutaneous treatment
  to assess the incidence of Major Adverse Cardiac and Cerebrovascular event (MACCE) individual components through 24 months
clinical improvement as assessed by Rutherford Class changes | within 6, 12 and 24 months vs baseline
  compare clinical improvement as assessed by Rutherford Class changes at 6, 12 and 24 months with respect to baseline

OTHER OUTCOMES:
rate of instrumental restenosis | within the first 24 months after percutaneous treatment
  the rate of instrumental restenosis as determined by duplex ultrasound Peak Systolic Velocity Ratio (PSVR) ≤ 2.4 post-index procedure and the rate of instrumental restenosis as determined by duplex ultrasound Peak Systolic Velocity Ratio (PSVR) ≤2 and ≤3.5 at 12 months (6, and 24 if available) or at unscheduled visit, as evaluated by an independent core lab
procedural success rate | at the end of percutaneous treatment
  rate of procedural success i.e. complete revascularization in the absence of peri-procedural complications
walking capacity and quality of life | whithin 6, 12 and 24 months post-procedure vs. baseline
  walking capacity as assessed by walking impairment questionnaire (WIQ) and quality of life (EQ5D questionnaire) at 6, 12 and 24 months post-procedure vs. baseline

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Micari, MD, Principal Investigator — Maria Eleonora Hospital, GVM Care & Research
Locations (6):
- Italy (6):
  - Anthea Hospital, Bari, Bari
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Città di Lecce Hospital, Lecce
  - Maria Eleonora Hospital, GVM Care & Research, Palermo
  - ICLAS Rapallo, Rapallo
  - Maria Pia Hospital, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Micari A, Vadala G, Castriota F, Liso A, Grattoni C, Russo P, Marchese A, Pantaleo P, Roscitano G, Cesana BM, Cremonesi A. 1-Year Results of Paclitaxel-Coated Balloons for Long Femoropopliteal Artery Disease: Evidence From the SFA-Long Study. JACC Cardiovasc Interv. 2016 May 9;9(9):950-6. doi: 10.1016/j.jcin.2016.02.014. PMID 27151609